CLINICAL TRIAL: NCT03011567
Title: A Randomized Controlled Trial on the Effects of NSAIDs on Postpartum Blood Pressure in Patients Hypertensive Disorders of Pregnancy
Brief Title: Hypertension In Postpartum Preeclampsia Study
Acronym: HIPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 663-15
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2020-08

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: Postpartum
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Severe HDP- NSAID (Experimental): This arm will be assigned a postpartum analgesic regimen with ibuprofen.
  Interventions: Drug: Ibuprofen
- Mild HDP- NSAID (Experimental): This arm will be assigned a postpartum analgesic regimen with ibuprofen.
  Interventions: Drug: Ibuprofen
- Severe HDP- No NSAID (Experimental): This arm will be assigned a postpartum analgesic regimen with acetaminophen.
  Interventions: Drug: Acetaminophen
- Mild HDP- No NSAID (Experimental): This arm will be assigned a postpartum analgesic regimen with acetaminophen.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Participants will receive acetaminophen for postpartum mild pain relief
  Other Names: Tylenol
  Arms: Mild HDP- No NSAID; Severe HDP- No NSAID
Drug: Ibuprofen — Participants will receive ibuprofen for postpartum mild pain relief
  Other Names: Motrin
  Arms: Mild HDP- NSAID; Severe HDP- NSAID

SUMMARY:
This study aims to evaluate whether NSAIDs (Non-steroidal antiinflammatory drugs) administered during the postpartum period influence blood pressure in women with hypertensive disorders of pregnancy. The study design is a prospective double blinded randomized control trial with participants randomized to receive postpartum analgesic regimens with and without NSAIDs.

DETAILED DESCRIPTION:
Non-steroidal antiinflammatory drugs (NSAIDs) are effective agents for the management of pain in the postpartum period. The addition of NSAIDs to post-cesarean analgesic regimen has been shown to improve post-cesarean pain and reduce opioid requirements. However, concern has been raised over use of NSAIDs in hypertensive pregnant patients, as recent evidence suggests the potential for increased blood pressure in patients with chronic hypertensive disorders receiving these agents. Notably, these studies were conducted on patients with longstanding chronic hypertension, which included males and non-pregnant females, and it is therefore unclear whether this recommendation is appropriate for patients with transient hypertensive disorders of pregnancy.

This protocol describes a randomized trial to evaluate whether NSAIDs influence blood pressure parameters in patients with hypertensive disorders of pregnancy. Patients with severe hypertensive disorders of pregnancy (Severe HDP) will be studied separately from women with mild hypertensive disorders of pregnancy (Mild HDP).

ELIGIBILITY:
Inclusion Criteria:

* Delivery occurred at equal to or greater than 24 0/7 weeks gestational age
* Patient receiving care with the Women's Perinatal Group (Maternal Fetal Medicine practice) or Obstetric Clinic resident services
* Diagnosis of a hypertensive disorder of pregnancy (HDP), including the following:
* Gestational hypertension
* Preeclampsia without severe features
* Preeclampsia with severe features
* Hemolysis, Elevated Liver Enzymes, Low Platelet (HELLP) Syndrome
* Eclampsia

Exclusion Criteria:

* Diagnosis of chronic hypertension or documentation of elevated blood pressures before 20 weeks gestational age.
* Severe hypertension: Patients with at least one severe blood pressure measurement (systolic >160mmHg or diastolic >105mmHg) prior to randomization
* Renal dysfunction (Serum creatinine measurement >1.3mg/dL during the current pregnancy)
* Low platelet count (recorded measurement <50,000 during hospital admission)
* Significant liver dysfunction (AST or ALT >500)
* Known sensitivities to ibuprofen or acetaminophen
* Use of therapeutic doses of anticoagulation (low dose anticoagulation used for routine prophylaxis of venous thromboembolism is acceptable)
* Postpartum hemorrhage requiring transfusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNulty, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (1):
- Miller Children and Women Hospital Long Beach, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Available on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Can be available on request
Access Criteria: Can be available on request

REFERENCES:
- [Derived] Penfield CA, McNulty JA, Oakes MC, Nageotte MP. Ibuprofen and Postpartum Blood Pressure in Women With Hypertensive Disorders of Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2019 Dec;134(6):1219-1226. doi: 10.1097/AOG.0000000000003553. PMID 31764732

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Hypertensive Disorders of Pregnancy (HDP)- NSAID; Mild Hypertensive Disorders of Pregnancy (HDP)- NSAID: This arm will be assigned a postpartum analgesic regimen with ibuprofen.
  Ibuprofen: Participants will receive ibuprofen for postpartum mild pain relief
- Severe Hypertensive Disorders of Pregnancy (HDP)- No NSAID; Mild Hypertensive Disorders of Pregnancy (HDP)- No NSAID: This arm will be assigned a postpartum analgesic regimen with acetaminophen.
  Acetaminophen: Participants will receive acetaminophen for postpartum mild pain relief
Period: Overall Study
Arm/Group | Severe Hypertensive Disorders of Pregnancy (HDP)- NSAID | Mild Hypertensive Disorders of Pregnancy (HDP)- NSAID | Severe Hypertensive Disorders of Pregnancy (HDP)- No NSAID | Mild Hypertensive Disorders of Pregnancy (HDP)- No NSAID
Started | 70 | 31 | 70 | 31
Randomized | 70 | 31 | 70 | 31
Completed | 70 | 31 | 70 | 30
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID | Total
Number analyzed (Participants) | 70 | 31 | 70 | 31 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 31 | 70 | 31 | 202
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.8) | 28 (6) | 29.2 (6.5) | 28 (5) | 28.5 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 31 | 70 | 31 | 202
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 12 | 46 | 11 | 106
  Not Hispanic or Latino | 33 | 19 | 24 | 20 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 5 | 3 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 7 | 10 | 5 | 38
  White | 47 | 18 | 54 | 20 | 139
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 70 | 31 | 70 | 31 | 202
Gestational age [Mean (Standard Deviation); unit: weeks] | 36.4 (4) | 37 (3) | 35.4 (3.7) | 38 (3) | 37 (1)

OUTCOME MEASURES:

1. Primary Outcome: Average Mean Arterial Blood Pressure- Mild Group
Description: Primary outcome for Hypertensive disorders of pregnancy-Mild Study Group
Time Frame: Averaged from all blood pressures measured through study completion, an average of 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Mild Hypertensive Disorders of Pregnancy- NSAID: This arm will be assigned a postpartum analgesic regimen with ibuprofen.
  Ibuprofen: Participants will receive ibuprofen for postpartum mild pain relief
- Mild Hypertensive Disorders of Pregnancy- No NSAID: This arm will be assigned a postpartum analgesic regimen with acetaminophen.
  Acetaminophen: Participants will receive acetaminophen for postpartum mild pain relief
Arm/Group | Mild Hypertensive Disorders of Pregnancy- NSAID | Mild Hypertensive Disorders of Pregnancy- No NSAID
Number analyzed (Participants) | 31 | 30
mmHg | 93 (8) | 93 (7)

2. Primary Outcome: Primary Outcome for Hypertensive Disorders of Pregnancy- Severe Study Group
Description: Proportion of participants with at least one episode of severe blood pressure postpartum (systolic >=160 or diastolic >=105mmHg) during inpatient postpartum hospitalization
Time Frame: Through study completion, an average of 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Severe Hypertensive Disorders of Pregnancy- NSAID: This arm will be assigned a postpartum analgesic regimen with ibuprofen.
  Ibuprofen: Participants will receive ibuprofen for postpartum mild pain relief
- Severe Hypertensive Disorders of Pregnancy- No NSAID: This arm will be assigned a postpartum analgesic regimen with acetaminophen.
  Acetaminophen: Participants will receive acetaminophen for postpartum mild pain relief
Arm/Group | Severe Hypertensive Disorders of Pregnancy- NSAID | Severe Hypertensive Disorders of Pregnancy- No NSAID
Number analyzed (Participants) | 70 | 70
Participants | 27 | 29

3. Secondary Outcome: Pain Control During Hospital Stay
Description: Wong-Baker Facial Grimace Pain Scale Scores During Inpatient Postpartum Hospital Stay Minimum 0, maximum 10. 10 means the highest level of pain
Time Frame: Through study completion, an average of 3 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID
Number analyzed (Participants) | 64 | 27 | 68 | 30
score on a scale | 6.1 (1.5) | 6.4 (1.4) | 5.6 (1.9) | 6.0 (1.0)

4. Secondary Outcome: Outpatient Blood Pressure Measurement
Description: Outpatient postpartum blood pressure measurement (represented in mean arterial pressure (MAP) within 6 weeks after discharge
Time Frame: 6 weeks after discharge from the hospital
Population: There was a large attrition in participants for this outpatient outcome
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Severe HDP-NSAID: These participants have severe antenatal hypertension and receive NSAIDs in the study medications
- Severe HDP-No NSAIDS: These participants have antenatal severe hypertension and do not receive NSAIDs in their study medications
Arm/Group | Mild HDP- NSAID | Mild HDP- No NSAID | Severe HDP-NSAID | Severe HDP-No NSAIDS
Number analyzed (Participants) | 8 | 9 | 17 | 20
mmHg | 99 [89.3 to 108.8] | 95 [84.5 to 104.5] | 97.8 [90.2 to 105.4] | 102.7 [96.9 to 108.4]

5. Secondary Outcome: Patient Satisfaction
Description: Number of patients reporting "High level of satisfaction with pain medications"
Time Frame: Through study completion, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID
Number analyzed (Participants) | 64 | 30 | 68 | 29
Participants | 58 | 22 | 65 | 22

6. Secondary Outcome: Length of Hospital Stay
Description: Length of Hospital Stay after delivery
Time Frame: Through study completion, an average of 3 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID
Number analyzed (Participants) | 70 | 23 | 70 | 23
days | 4.3 [1.9 to 6.7] | 2.0 [1.71 to 2.3] | 3.7 [2.7 to 4.7] | 1.8 [1.56 to 1.95]

7. Secondary Outcome: Diuresis
Description: Achievement of average 200ml/hour for 4 consecutive hours
Time Frame: Through study completion, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID
Number analyzed (Participants) | 70 | 31 | 70 | 30
Participants | 45 | 19 | 46 | 23

8. Secondary Outcome: Average Mean Arterial Blood Pressures During Hospital Stay
Time Frame: Averaged from all blood pressures measured through study completion, an average of 3 days
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Severe Hypertensive Disorders of Pregnancy- NSAID | Severe Hypertensive Disorders of Pregnancy- No NSAID
Number analyzed (Participants) | 70 | 70
mmHG | 95.7 (8.2) | 95.9 (9.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study enrollment until 6 weeks postpartum.
Arm/Group | Severe HDP- NSAID | Mild HDP- NSAID | Severe HDP- No NSAID | Mild HDP- No NSAID
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/31 | 0/70 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/31 | 0/70 | 0/30
Other Adverse Events (participants affected / at risk) | 0/70 | 0/31 | 0/70 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03011567/Prot_SAP_000.pdf